CLINICAL TRIAL: NCT04570826
Title: EFFECTS OF A MEDITATION PROGRAM ON THE QUALITY OF LIFE IN HIGH-BURDEN INFORMAL CAREGIVERS
Brief Title: A MEDITATION PROGRAM IN HIGH-BURDEN INFORMAL CAREGIVERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consuelo Lourdes Díaz Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Consuelo Lourdes Díaz Rodríguez, Sponsor-Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2020-08-30; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Caregivers Burnout
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Intervention Model Description: A meditation master practitioner with at least 10 years of experience implemented in the Faculty of Health Sciences of the University of Granada a FAM program during four weeks, two sessions per week, each Friday. The caregiver attendance to two continues sessions during a total of four hours, two hours per session with thirty minutes of rest between both of them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation program (Experimental): The experimental group participated in the Meditation program during one month, eight sessions with a total of sixteen hours.
  Interventions: Other: Meditation.
- Scientific descriptions about meditation (Active Comparator): The control group received scientific descriptions about meditation.
  Interventions: Other: Scientific descriptions about meditation.

INTERVENTIONS:
Other: Meditation. — The caregivers received eight sessions lasting each one two hours with the following sequence: before each practical exercises they always received 15 minutes about scientific theoretical evidence explaining the importance of doing them: to get a comfortable posture they received 25 minutes of mobility, flexibility, balance, strength and endurance exercises. To increase lung capacity, 25 minutes of costal, diaphragmatic and clavicular breathing exercises. Finally, to have an open attitude without distractions or judging they practiced 25 minutes of body awareness exercise observing sensations, thoughts and perceptions with gratitude and compassion.
  Arms: Meditation program
Other: Scientific descriptions about meditation. — The control group received scientific descriptions about meditation.
  Arms: Scientific descriptions about meditation

SUMMARY:
The aim of the present study was to investigate in high burden caregivers the effects of a face-to-face meditation program during four weeks (16 hours) on physiological parameters, psychological state and vagal nerve activity comparing with a control group.

DETAILED DESCRIPTION:
A non-randomized repeated-measures controlled clinical trial was conducted with convenience allocation of participants into intervention (n = 18) or control group (n = 17). Due to ethical reasons, it was not possible to randomize the patients.

The investigators invited from different associations in Granada city and its province through word and mouth or by telephone to 45 volunteer informal caregivers. 40 of them enrolled in this study but only 37 finalized the program, 24.3% male and 75.7% female with a mean (SD) age of 44.03 (7.30) years. The people that have previous experience in mind body practices or cardiovascular diseases were excluded. All the caregivers received information about the study and informed consent was obtained from all participants. This study was approved by the CEI-GR (C-9) ethics committee and followed the principles of the Declaration of Helsinki. Convenience sampling was used to assign caregivers to the control or experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* People who care for a dependent family member or close relative and live with him/her in the same home for at least two years with a caregiver burden of more than 55 points in Zarit Burden Scale.

Exclusion Criteria:

* People that have previous experience in mind body practices or cardiovascular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Happiness on the Lima happiness questionnaire after 1 month | Baseline and after 1 month
  Lima happiness questionnaire: Validated self-administered questionnaire consisting of 27 items, integrated into 4 subscales (Positive sense of life, Satisfaction with life, Personal fulfillment and Joy of life), which refer to the level of happiness or satisfaction that the person has with respect to his life.
  The respondent may be: (1) Strongly agree, (2) Agree, (3) Neither agree nor disagree, (4) Disagree or (5) Strongly disagree, with any question that arises. According to the total score there are 5 levels of happiness: from 27-87: very low happiness, 88-95: low, 96-110: medium, 111-118: high, 119-135: very high.
Change from Baseline in Anxiety and Depression on the Hospital Anxiety and Depression Scale (HADS) after 1 month | Baseline and after 1 month
  Validated self-administered instrument for outpatients that advises on the possible presence of anxiety and depression in any non-psychiatric medical consultation. Describe how the patient feels affective and emotionally during the last week.
  It has 14 items, 7 for each subscale with a scale similar to four points (from 0 to 3). Lower scores reflect better outcomes.
Change from Baseline in Heart rate and Heart rate variability after 1 month | Baseline and after 1 month
  We measured short-term HRV using an accepted method in order to assess the cardiovascular balance (Kappussami 2020). We asked participants to lie in a supine position for 10 min of rest with normal breathing (following a metronome at 0.2 Hz) and no external stimulation in a quiet room with a temperature of 22-25 °C.
Change from Baseline in Blood pressure/heart rate after 1 month | Baseline and after 1 month
  We measured blood pressure and heart rate before and after the treatment session using an Omron HEM-7320-Z validated automatic oscillometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Lourdes Díaz Rodríguez, Granada, Spain